CLINICAL TRIAL: NCT01729611
Title: Endothelial Function in Patients With Scleroderma or Cirrhosis With and Without Pulmonary Hypertension
Status: Completed | Type: Observational
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, Adriano Tonelli, Staff Physician, The Cleveland Clinic
Other Study IDs: Tonella1
Record Dates: First submitted 2012-11-15; First posted 2012-11-20 (Estimated); Last update posted 2021-04-02 (Actual); Status verified 2021-04

CONDITIONS: Pulmonary Hypertension
Keywords: Scleroderma; Cirrhosis
MeSH Terms: conditions — Hypertension, Pulmonary; Scleroderma, Diffuse; Fibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Scleroderma: 60 patients with scleroderma - 30 with and 30 without Pulmonary Arterial Hypertension
- Cirrhosis: 60 patients with cirrhosis - 30 with and 30 without Pulmonary Arteria Hypertension

SUMMARY:
Pulmonary arterial hypertension (PAH) is a condition characterized by an increased pulmonary vascular resistance that can lead to right heart failure and death. Several diseases are known etiologies of PAH including scleroderma and cirrhosis. The presence of PAH in the context of systemic sclerosis or cirrhosis has a dramatic impact on prognosis and survival of the connective tissue or liver disease.

Despite advances in the diagnosis of PAH, echocardiography remains a necessary test for screening PAH in patients with scleroderma or cirrhosis. However, echocardiography is less than ideal for diagnosing PAH and predicting treatment response. Thus, there is a pressing need to identify methodologies that can accurately and non-invasively recognize the presence of PAH in patients with scleroderma and cirrhosis.

Hypothesis:

1. To measure endothelial function and exhaled gases in patients with scleroderma and cirrhosis. To assess whether they correlate with the presence or the development of PAH.
2. The degree of local (forearm) capillary vasodilation during treprostinil iontophoresis identifies patients who will develop PAH and in those already diagnosed PAH predicts response to PAH-specific therapies.

DETAILED DESCRIPTION:
Patients with scleroderma are known to have endothelial dysfunction and limited data suggested an association between the degree of endothelial function in scleroderma and the presence of PAH. However, these data is preliminary and has not been used to predict response to PAH-specific therapy or the development of PAH. We will test patients with cirrhosis because they tend to have PAH in the context of a hyperdynamic instead of a hypodynamic state as observed in scleroderma and PAH.

Aims:

1. To measure endothelial function and exhaled gases in patients with scleroderma or cirrhosis to assess whether they correlate with the presence or the development of PAH.
2. To evaluate the degree of endothelial response to local treprostinil iontophoresis and determine if this test can predict the development of pulmonary hypertension or response to PAH-specific therapies.

ELIGIBILITY:
Inclusion Criteria:

* Patients with scleroderma or cirrhosis.

Exclusion Criteria:

* Exclusion criteria include individuals younger than 16, etiologies of PAH other than scleroderma or cirrhosis.

Ages: 17 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with scleroderma or cirrhosis. These patients may or may not have known PAH or be on treatment of this condition.
Sampling Method: Non-Probability Sample
Enrollment: 119 (Actual)
Dates: Start 2013-12 (Actual); Primary Completion 2021-03 (Actual); Study Completion 2021-04 (Actual)

PRIMARY OUTCOMES:
Base Line | up to 3 months
  Baseline characteristics in patients with and without PAH will be compared using parametric (t-test) and non parametric (Mann-Whitney) tests for continuous data and Chi-square for categorical data.

CONTACTS AND LOCATIONS:
Overall Officials: Adriano Tonelli, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States